CLINICAL TRIAL: NCT03419520
Title: Detection of Genetic Polymorphisms Associated With Obesity and Its Complications in Schoolchildren Within the Madrid Community, and Evaluation of Health Actions for Reducing the Risk
Brief Title: GENYAL Study to Childhood Obesity Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IMDEA Food (Other)
Responsible Party: Principal Investigator, Viviana Loria Kohen, Senior Nutritionist, PhD in Medicine. Researcher and Group leader of the Nutrition and Clinical Trials Unit, IMDEA Food
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IMD PI0024
Record Dates: First submitted 2018-01-19; First posted 2018-02-05 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Childhood Onset Obesity
Keywords: Schoolchildren; Overweight; Obesity; Polymorphisms; Genetics; Nutritional counseling; Healthy strategies
MeSH Terms: conditions — Pediatric Obesity; Overweight; Obesity | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: The present study is an observational and long-term intervention study. There is an initial evaluation carried out on all children involved in the study at 1st and 2nd grades and it is going to be followed by 3 monitoring actions in the following years where the progression of anthropometric measurements and dietary habits are going to be studied. Besides, the intervention group is going to receive nutritional education aimed to reduce the risk of developing obesity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Schools receive healthy actions aimed to reduce the risk of developing obesity, along the study
  Interventions: Behavioral: Nutritional counseling
- Control group (No Intervention): Schools monitored along the study but won't receive any healthy action.

INTERVENTIONS:
Behavioral: Nutritional counseling — Schoolchildren, parents and teachers from intervention schools, will regularly receive nutrition and healthy lifestyle guidelines performed by nutritionists. Moreover, workshops aimed to reinforce the healthy habits will also be held along the study.
  Arms: Intervention group

SUMMARY:
Obesity is a multifactorial, complex, chronic disease of special concern. It is originated as an interaction between genetic predisposition and environmental factors. Thus, knowledge of gene-diet interactions is especially important. However, most studies analyzing the efficacy of diet on body weight have not considered the genetic variability among the population.

Childhood and adolescence are critical periods in the development of obesity. This is because, on one hand, during infancy dietary patterns are being implemented. Moreover, it has been described that around the age of 6 it occurs the adiposity rebound, which consists in the increase in body mass index (BMI) that occurs after reaching a lowest point in infancy. It is believed that an early adiposity rebound is associated with a higher risk of developing obesity in the following years. The prevalence of overweight and obese children is increasing every year. Specifically, according to the World Health Organization (WHO) the number of overweight or obese children aged 0 to 5 years, increased from 32 million globally in 1990 to 41 million in 2016. Regarding Spanish children, they are amongst the highest levels of overweight and obesity in Europe. Precisely, in 2015 the Spanish Agency for Consumer Affairs, Food Safety and Nutrition reported 23.2 % overweight and 18.1 % obese Spanish children, according to the ALADINO study.

Considering the previous elaboration, we hypothesized that an early identification of SNPs associated with obesity will improve the strategies applied for its prevention. Moreover, an adequate nutritional counseling and a healthy lifestyle implementation during childhood will contribute to a higher quality of life in the adulthood.

Thus, schools from the Madrid Community agreeing to participate in the study will be randomly assigned to either control or intervention groups. Then, an initial evaluation where 26 SNPs associated with obesity and its related comorbidities will be carried out in all children involved in the study, in addition to anthropometric, blood pressure measurements, and physical activity and dietary patterns evaluation. Then, each group will be divided in two according to the genetic risk (high vs low) for presenting obesity and its related comorbidities. The initial evaluation was performed on all children at 1st and 2nd grades and it is going to be followed by 3 monitoring actions in the following years where the progression of anthropometric measurements and dietary habits are going to be studied. Besides, the intervention schools are going to receive healthy actions along the study aimed to reduce the risk of developing obesity.

ELIGIBILITY:
Inclusion Criteria:

Children at 1st and 2nd grades from schools of the Madrid Community that have accepted to participate in the study, whose parents have approved and signed the informed consent.

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 221 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Changes in the percentage of children with a diagnosis of obesity | There will be an initial assessment followed by 2 evaluations in the two consecutive years and a third and final evaluation 4 years after the initial assessment.
  The International Obesity Task Force classification will be used to the diagnosis of obesity

SECONDARY OUTCOMES:
Changes in energy intake | There will be an initial assessment followed by 2 evaluations in the two consecutive years and a third and final evaluation 4 years after the initial assessment.
  A 48h food record and the DIAL (Alce Ingenieria) software will be used to evaluate the energy intake (Kcal) of the studied population
Changes in body fat mass percentage | There will be an initial assessment followed by 2 evaluations in the two consecutive years and a third and final evaluation 4 years after the initial assessment.
  The fat mass percentage will be measured using the Body Composition Monitor (BF511- OMRON HEALTHCARE UK, LT, Kyoto, Japan)
Physical activity | There will be an initial assessment followed by 2 evaluations in the two consecutive years and a third and final evaluation 4 years after the initial assessment.
  A 24h physical activity questionnaire and the Institute of Medicine of the National Academies classification will be used to measure the physical activity level
Genetic predisposition to develop obesity | There will be an initial assessment at the beginning of the study
  A total of 26 SNPs related to obesity development will be analysed using saliva samples and the QuantStudio™ 12K Flex (Life Technologies) equipment. (Machine learning predictive modeling)

CONTACTS AND LOCATIONS:
Overall Officials: Guilerrmo Reglero, Professor, Study Director — IMDEA Food; Ana Ramirez-de Molina, PhD, Study Director — IMDEA Food
Locations (1):
- IMDEA-Food, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Marcos-Pasero H, Aguilar-Aguilar E, de la Iglesia R, Espinosa-Salinas I, Molina S, Colmenarejo G, Martinez JA, Ramirez de Molina A, Reglero G, Loria-Kohen V. "GENYAL" Study to Childhood Obesity Prevention: Methodology and Preliminary Results. Front Nutr. 2022 Mar 8;9:777384. doi: 10.3389/fnut.2022.777384. eCollection 2022. PMID 35350411
- [Derived] Marcos-Pasero H, Aguilar-Aguilar E, de la Iglesia R, Espinosa-Salinas I, Gomez-Patino M, Colmenarejo G, de Molina AR, Reglero G, Loria-Kohen V. Association of calcium and dairy product consumption with childhood obesity and the presence of a Brain Derived Neurotropic Factor-Antisense (BDNF-AS) polymorphism. Clin Nutr. 2019 Dec;38(6):2616-2622. doi: 10.1016/j.clnu.2018.11.005. Epub 2018 Nov 20. PMID 30501916